CLINICAL TRIAL: NCT02300948
Title: Optimizing Periconceptional and Prenatal Folic Acid Supplementation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Duchesnay Inc. (Industry)
Responsible Party: Principal Investigator, Gideon Koren, Director of MotherRisk Program, Clinical Pharmacology and Toxicology, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1000009554
Record Dates: First submitted 2014-11-21; First posted 2014-11-25 (Estimated); Last update posted 2014-11-25 (Estimated); Status verified 2014-11

CONDITIONS: Pregnancy
Keywords: Pregnancy; Perinatal Vitamins; folate
MeSH Terms: interventions — Folic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PregVit-Folic 5®-5 mg folic acid (Experimental): Prenatal multivitamin-mineral supplement called PregVit-folic 5® contains 5 mg of folic acid. All other vitamin and mineral doses are identical between the 2 supplements, except for folic acid. Both supplements are taken as 2 tablets daily, one tablet in the morning (am) and one tablet in the evening (pm). Both multivitamins are appropriate for periconceptional, prenatal, and post-partum supplementation.
  Interventions: Drug: PregVit-folic 5® contains 5 mg of folic acid
- PregVit®-1.1 mg folic acid (Active Comparator): Prenatal multivitamin-mineral supplement called PregVit® contains 1.1 mg of folic acid. All other vitamin and mineral doses are identical between the 2 supplements, except for folic acid. Both supplements are taken as 2 tablets daily, one tablet in the morning (am) and one tablet in the evening (pm). Both multivitamins are appropriate for periconceptional, prenatal, and post-partum supplementation.
  Interventions: Drug: PregVit® contains 1.1 mg of folic acid

INTERVENTIONS:
Drug: PregVit® contains 1.1 mg of folic acid — Participants are randomly allocated to one of two groups: PregVit-Folic 5® (group1) contains 5 mg folic acid or PregVit® (group 2) contains 1.1 mg folic acid.Both supplements are taken as 2 tablets daily, one tablet in the morning (am) and one tablet in the evening (pm). Both multivitamins are appropriate for periconceptional, prenatal, and post-partum supplementation. The total volume of blood that will be taken is approximately 20 mL (4 teaspoons). Each appointment will be scheduled according to when participants are available. To monitor adherence, the PregVit-Folic 5® blister packs should be returned among with a diary of pill intake (will be provided). To document dietary folate, telephone interviews regarding the diet will be conducted.
  Other Names: Pregvit®
  Arms: PregVit®-1.1 mg folic acid
Drug: PregVit-folic 5® contains 5 mg of folic acid — Participants are randomly allocated to one of two groups: PregVit-Folic 5® (group1) contains 5 mg folic acid or PregVit® (group 2) contains 1.1 mg folic acid.Both supplements are taken as 2 tablets daily, one tablet in the morning (am) and one tablet in the evening (pm). Both multivitamins are appropriate for periconceptional, prenatal, and post-partum supplementation. The total volume of blood that will be taken is approximately 20 mL (4 teaspoons). Each appointment will be scheduled according to when participants are available. To monitor adherence, the PregVit-Folic 5® blister packs should be returned among with a diary of pill intake (will be provided). To document dietary folate, telephone interviews regarding the diet will be conducted.
  Other Names: PregVit Folic 5®
  Arms: PregVit-Folic 5®-5 mg folic acid

SUMMARY:
There are three objectives in this study:

1. To assess the serum folate pharmacokinetics of ingesting a single dose of PregVit-Folic5® versus a single dose of PregVit® (a multivitamin containing 1.1 mg folic acid)
2. To assess the steady-state red blood cell (RBC) and serum folate concentrations achieved in non-pregnant, fertile women who supplement daily with PregVit-Folic5® versus PregVit®
3. To assess the steady-state RBC and serum folate concentrations achieved before and during pregnancy in women planning a pregnancy or early in pregnancy (<6 weeks gestation) who supplement daily with PregVit-Folic5® versus PregVit®.

DETAILED DESCRIPTION:
A prospective, randomized, 2-arm, interventional study involving women of child-bearing age will compare the folate status and pharmacokinetics of PregVit-Folic5® and PregVit®.

Some women of childbearing age, particularly those who do not practice multivitamin supplementation, may have inadequate intake and blood concentrations of vitamins and minerals, including those micronutrients which are important in pregnancy. Folic acid is one of the important vitamins in pregnancy which can be obtained from folate-rich foods, folic acid-fortified foods, and multivitamins. It is important to examine the folate status of fertile women, who do not usually practice multivitamin supplementation, before and after they implement folic acid containing-multivitamin supplementation.

The investigators wish to measure red blood cell and serum folate concentrations among women who are healthy and/or childbearing age, those planning a pregnancy or early in pregnancy (< 6 weeks gestation) and who do not practice multivitamin supplementation. The investigators would like to measure and compare folate levels among women before and after implementing multivitamin supplementation with either PregVit® or PregVit-Folic 5®. This may be important information for planning or pregnant women who need folic acid, which has been shown to reduce the risk of neural tube defects and potentially other malformations as well.

The Study hypotheses are as follows:

1. The serum folate concentration from ingesting PregVit-folic 5® (5 mg folic acid) will be 4-5 fold larger compared to that of PregVit® (1.1 mg folic acid).
2. Non-pregnant women of childbearing age who supplement daily with PregVit-folic 5® will invariably and optimally achieve and maintain maximum protective blood folate levels (i.e. ≥900 nM red blood cell folate) against NTDs.
3. Women planning a pregnancy or early in pregnancy (<6 weeks gestation) who supplement daily with PregVit-folic 5® will invariably and optimally achieve and maintain maximum protective blood folate levels (i.e. ≥ 900 nM red blood cell folate) against NTDs before and during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Any healthy, non-pregnant, fertile woman between 18 and 45 years of age.(Part 1 and 2)
* Have not taken multivitamins or folic acid supplements in the past 6 months. (Part 1 and 2)
* Healthy women between 18 to 45 years of age.(For Part 3)
* Planning a pregnancy, or within the first 2 weeks of missing a menstrual period, or within the first 6 weeks of pregnancy.(Part 3)
* Have not taken multivitamins or folic acid supplements in the past 6 months.(Part 3)

Exclusion Criteria:

* Have hypersensitivities to the ingredients in PregVit-folic 5® or PregVit®. (Part 1, 2 and 3)
* Have chronic medical conditions (i.e. hypertension, diabetes, epilepsy, irritable bowel syndrome, hypo/hyper-thyroidism, depression). (Part 1, 2 and 3)
* Chronic use (i.e. long-term, specifically prescribed dose) of oral medications (i.e. oral contraceptives, anticonvulsants, antibiotics, antidepressants).(Part 1, 2 and 3)
* Have a family history or previous pregnancy affected by NTDs.(Part 1, 2 and 3)
* Do not agree to the protocol.(Part 1, 2 and 3)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 83 (Actual)
Dates: Start 2006-12; Primary Completion 2013-02 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
The serum folate pharmacokinetics in healthy, non-pregnant women of childbearing age who ingest a single evening dose of PregVit-folic 5® (5 mg folic acid) versus a single evening dose of PregVit® (1.1 mg folic acid). | 1 day
  For the single dose study, extensive blood sampling was conducted over 12 hours.
The steady-state red blood cell and serum folate levels achieved in healthy, non-pregnant women of childbearing age who supplement daily for 30 weeks with PregVit-folic 5® versus PregVit®. | 6 days
  The first clinic visit will be to draw blood (5 mL) to measure baseline red blood cell folate, plasma folate, and vitamin B12 concentrations (after a 6 hour fast). Then blood samples will be drawn at weeks 2, 4, and 6 of study participation to measure RBC and plasma folate levels to determine what peak level is achieved and the time required to achieve the peak (or achieve RBC folate concentration of 900 nM or greater). As supplementation continues, RBC and plasma folate levels will be measured again at 12 and 30 weeks of participation.
The steady-state periconceptional and gestational red blood cell and serum folate levels in women planning a pregnancy or early in pregnancy (<6 weeks gestation) who supplement daily with PregVit-folic 5® versus PregVit®. | 4 days
  For the multiple dose study, blood sampling was conducted as follows:
  The first clinic visit will be to draw blood (5 mL) to measure baseline red blood cell folate, plasma folate, and vitamin B12 concentrations (after a 6 hour fast). Return to research site at 6 weeks gestation to draw one blood sample. Pick up next supply of multivitamins (hospital pharmacy).
  Return to research site at 12 weeks gestation to draw one blood sample. Pick up next supply of multivitamins (hospital pharmacy).
  Return to research site at 30 weeks gestation to draw last blood sample.

CONTACTS AND LOCATIONS:
Overall Officials: Gideon Koren, MD, Principal Investigator — The Hospital for Sick Children, Toronto Canada
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada